CLINICAL TRIAL: NCT03118440
Title: Multi-center, Randomized, Controlled Trial to Compare Feasibility, Safety and Efficacy of Zero-Fluoroscopic Navigation With Conventional Fluoroscopic Navigation for Single-chamber Pacemaker Implantation
Brief Title: Zero-fluoroscopic Navigation Versus Conventional Fluoroscopic Navigation for Single-chamber Pacemaker Implantation
Acronym: ZF-PMSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other); Xinyang Central Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Guangdong Provincial People's Hospital (Other); Wuhan Asia Heart Hospital (Other); Shenzhen Sun Yat-sen Cardiovascular Hospital (Other); Ningbo No. 1 Hospital (Other)
Responsible Party: Principal Investigator, Yan Wang, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJHCDC-ZF-PMSC-20130101
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Sick Sinus Syndrome; Complete Atrioventricular Block; High Degree Second Degree Atrioventricular Block; Bradycardia
Keywords: Fluoroscopy; Pacemaker; Three dimensional; Radiation; Imaging
MeSH Terms: conditions — Sick Sinus Syndrome; Bradycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero-fluoroscopy implantation (Experimental): Pacemaker implantation performed for all patients in this group with zero-fluoroscopy 3D navigation.
  Interventions: Procedure: zero-fluoroscopy 3D navigation
- Conventional fluoroscopy implantation (Active Comparator): Pacemaker implantation performed for all patients with conventional x-ray navigation.
  Interventions: Procedure: conventional x-ray navigation

INTERVENTIONS:
Procedure: zero-fluoroscopy 3D navigation — Pacemaker implantation will be performed without fluoroscopy using 3D navigation systems.
  Other Names: non-fluoroscopy 3D navigation
  Arms: Zero-fluoroscopy implantation
Procedure: conventional x-ray navigation — Pacemaker implantation will be performed with fluoroscopy using conventional X-ray navigation.
  Other Names: fluoroscopy navigation
  Arms: Conventional fluoroscopy implantation

SUMMARY:
This study is intended to compare the feasibility, safety and efficacy of Ensite-NavX zero-fluoroscopic navigation system to conventional fluoroscopic X-ray approach as to performing single-chamber pacemaker implantation.

DETAILED DESCRIPTION:
Permanent pacemaker is a well-established treatment to treat patients with a wide range of heart rhythm disturbances.

Fluoroscopy is the imaging modality routinely used for cardiac device implantation and electrophysiological procedures.Due to the rising concern regarding the harmful effects of radiation exposure to both the patients and operation staffs, novel 3D mapping systems have been developed and implemented in electrophysiological procedure for the navigation of catheters inside the heart chambers.

Ensite NavX system can be used for cardiac imaging as a reliable and safe zero-fluoroscopy approach for implantation of single- or dual-chamber permanent pacemaker in patients. Our method offered a choice for some special population of patient in whom radiation exposure need to be avoided or in the extreme circumstances when the X-ray machine is out-of-order.

ELIGIBILITY:
Inclusion Criteria:

* Sick Sinus Syndrome
* complete Atrioventricular Block
* high degree second Degree Atrioventricular Block
* Bradycardia

Exclusion Criteria:

* pacemaker replacement
* severe structural l cardiac malformations
* severe cardiac enlargement
* venous malformations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Success rate | 3 months

SECONDARY OUTCOMES:
Total procedure time | during procedure
Fluoroscopy time | during procedure
Complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller DL, Balter S, Schueler BA, Wagner LK, Strauss KJ, Vano E. Clinical radiation management for fluoroscopically guided interventional procedures. Radiology. 2010 Nov;257(2):321-32. doi: 10.1148/radiol.10091269. PMID 20959547
- [Background] Ventura R, Rostock T, Klemm HU, Lutomsky B, Demir C, Weiss C, Meinertz T, Willems S. Catheter ablation of common-type atrial flutter guided by three-dimensional right atrial geometry reconstruction and catheter tracking using cutaneous patches: a randomized prospective study. J Cardiovasc Electrophysiol. 2004 Oct;15(10):1157-61. doi: 10.1046/j.1540-8167.2004.04064.x. PMID 15485440
- [Background] Gepstein L, Hayam G, Ben-Haim SA. A novel method for nonfluoroscopic catheter-based electroanatomical mapping of the heart. In vitro and in vivo accuracy results. Circulation. 1997 Mar 18;95(6):1611-22. doi: 10.1161/01.cir.95.6.1611. PMID 9118532
- [Background] Lemery R. Interventional electrophysiology at the crossroads: cardiac mapping, ablation and pacing without fluoroscopy. J Cardiovasc Electrophysiol. 2012 Oct;23(10):1087-91. doi: 10.1111/j.1540-8167.2012.02373.x. Epub 2012 Aug 6. No abstract available. PMID 22882722
- [Background] Richter S, Doring M, Gaspar T, John S, Rolf S, Sommer P, Hindricks G, Piorkowski C. Cardiac resynchronization therapy device implantation using a new sensor-based navigation system: results from the first human use study. Circ Arrhythm Electrophysiol. 2013 Oct;6(5):917-23. doi: 10.1161/CIRCEP.113.000066. Epub 2013 Sep 3. PMID 24002003
- [Background] Wittkampf FH, Wever EF, Derksen R, Wilde AA, Ramanna H, Hauer RN, Robles de Medina EO. LocaLisa: new technique for real-time 3-dimensional localization of regular intracardiac electrodes. Circulation. 1999 Mar 16;99(10):1312-7. doi: 10.1161/01.cir.99.10.1312. PMID 10077514
- [Background] Schreieck J, Ndrepepa G, Zrenner B, Schneider MA, Weyerbrock S, Dong J, Schmitt C. Radiofrequency ablation of cardiac arrhythmias using a three-dimensional real-time position management and mapping system. Pacing Clin Electrophysiol. 2002 Dec;25(12):1699-707. doi: 10.1046/j.1460-9592.2002.01699.x. PMID 12520670